CLINICAL TRIAL: NCT03529565
Title: The Role of Histamine in Breast Cancer Bone Pain
Brief Title: Histamine and Bone Pain Association in Participants With Breast Cancer Metastatic in the Bone
Status: Terminated | Type: Observational
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00048455; NCI-2018-00277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 02217 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-05-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Bone Pain; Breast Carcinoma Metastatic in the Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Participants undergo collection of blood samples for histamine level analysis via ELISA.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies histamine and bone pain association in participants with breast cancer that has spread to the bone. Studying histamine levels in samples of blood from participants with breast cancer in the laboratory may help doctors learn more about reducing cancer bone pain and preventing further bone metastasis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate levels of histamine in plasma with pain scores in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy.

SECONDARY OBJECTIVES:

I. To perform exploratory studies with additional markers not mentioned, including calcitonin gene-related peptide (CGRP), stem cell factor (SCF), angiotensin II (Ang II) substance P, angiotensin 1-7 (Ang1-7), may be performed at the investigator's discretion.

II. To perform next generation ribonucleic acid (RNA) sequences using the whole blood to determine whether histamine system is involved in the development of cancer-induced bone pain (CIBP).

III. To assess the impact of pain response after radiotherapy on bone structural properties such as bone mineral density and cortical thickness, and patient quality of life, physical and psychological function.

OUTLINE:

Participants undergo collection of blood samples for histamine level analysis via enzyme-linked immunosorbent assay (ELISA).

After completion of study, participants are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with radiographic evidence of bone metastases (by plain film, computed tomography [CT], magnetic resonance imaging [MRI], positron emission tomography [PET] or bone scan) within 8 weeks of registration

  * Weight bearing sites: pelvis (excluding pubis), femur, sacrum and/or sacroiliac joints, tibia, up to 5 consecutive cervical, thoracic or lumbar vertebral bodies, lumbosacral spine
  * Non-weight bearing sites: up to 3 consecutive ribs, humerus, fibula, radius +/- ulna, clavicle, sternum, scapula, pubis
* Patients with and without pain related to the radiographically documented metastases are eligible for study
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Pregnant women will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with breast cancer with radiographic evidence of bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Plasma histamine levels | Up to 6 months
  To correlate levels of histamine in plasma with pain scores (3 groups) in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy, analysis of variance (ANOVA) will be used. The histamine levels will be transformed to satisfy the conditional normality assumption if needed. Linear regression models will be used to relate histamine levels (outcome variable) with the pain groups (covariate of interest).

SECONDARY OUTCOMES:
Calcitonin gene-related peptide (CGRP) | Up to 6 months
  Levels of CGRP will be collected. Statistical analysis will correlate CGRP with pain scores (3 groups) in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy, ANOVA will be used.
Stem cell factor (SCF) | Up to 6 months
  Levels of SCF will be collected. Statistical analysis will correlate SCF with pain scores (3 groups) in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy, ANOVA will be used.
angiotensin II (Ang II) Substance P | Up to 6 months
  Levels of Ang II will be collected. Statistical analysis will correlate Ang II with pain scores (3 groups) in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy, ANOVA will be used.
angiotensin 1-7 (Ang1-7) levels | Up to 6 months
  Levels of Ang 1-7 will be collected. Statistical analysis will correlate Ang 1-7 with pain scores (3 groups) in patients with bone metastases from breast cancer that have or have not been treated with palliative radiotherapy, ANOVA will be used.
Histamine system involvement | Up to 6 months
  Will perform next generation ribonucleic acid (RNA) sequences using whole blood to determine whether histamine system is involved in the development of cancer-induced bone pain (CIBP).
Change in bone structural properties | Baseline up to 1 month
  The thickness of the cortical bone within the irradiated volume will be measured.
Change in patient quality of life | Baseline up to 1 month
  The change in patient quality of life will be assessed by the visual analogue scale (VAS) pain scale. The total score range is 0-10 with higher scores denoting worse outcomes.
Change in physical and psychological function | Baseline up to 1 month
  To be measured using the EORTC QLQ-BM22 quality of life questionnaire. It's divided into two categories, giving a single value: symptoms and functions. A high score indicates a high level of symptoms and a high level of functioning. The score range is 22-88.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Brown, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03529565/ICF_000.pdf